CLINICAL TRIAL: NCT00643851
Title: A Multicenter, Randomized, Double-Blind, Active Controlled, Parallel Group, Phase 3 Trial to Evaluate the Safety and Efficacy of Dapagliflozin in Combination With Metformin as Initial Therapy as Compared With Dapagliflozin Monotherapy and Metformin Monotherapy in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control
Brief Title: An Efficacy & Safety Study of BMS-512148 in Combination With Metformin Extended Release Tablets
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB102-021
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): Dapagliflozin (5 mg) + Metformin XR (up to 2000 mg)
  Interventions: Drug: Dapagliflozin; Drug: Metformin XR
- Arm 2 (Experimental): Dapagliflozin (5 mg)
  Interventions: Drug: Dapagliflozin
- Arm 3 (Active Comparator): Metformin XR (500 mg up to 2000 mg)
  Interventions: Drug: Metformin XR

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, Once daily, 24 weeks
  Other Names: BMS-512148
  Arms: Arm 1; Arm 2
Drug: Metformin XR — Tablets, Oral, Once daily, 24 weeks
  Arms: Arm 1; Arm 3

SUMMARY:
The purpose of this clinical research study is to learn if initiating treatment with BMS-51248 (Dapagliflozin) in combination with metformin XR can improve diabetes control in patients with Type 2 Diabetes who do not receive any pharmacological treatment for diabetes, when compared to initial treatment with monotherapy dapagliflozin or metformin XR. The safety of this treatment will also be studied

ELIGIBILITY:
Inclusion Criteria:

* Males & females, 18-77 years old inclusive, with type 2 diabetes and with inadequate glycemic control
* Drug naive or treated with anti-diabetic medication for < 24 weeks since original diagnosis
* C-peptide ≥ 1.0 ng/mL
* Body Mass Index ≤ 45.0 kg/m
* Serum creatinine < 1.50 mg/dL for men or < 1.40 mg/dL for women

Exclusion Criteria:

* AST and/or ALT >3.0 times the upper limit of normal (ULN)
* Serum total bilirubin > 2.0 mg/dL
* Creatine kinase > 3X the upper limit of normal (ULN)
* Symptoms of severely uncontrolled diabetes
* Currently unstable or serious cardiovascular, renal, hepatic, hematological, oncological, endocrine, psychiatric or rheumatic diseases

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 994 (Actual)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (89):
- United States (44):
  - Greystone Medical Research, Llc, Birmingham, Alabama
  - Winston Technology Research, Llc, Haleyville, Alabama
  - Clinical Research Advantage, Inc., Tempe, Arizona
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Southland Clinical Research Center, Inc., Fountain Valley, California
  - Valley Research, Fresno, California
  - Central Florida Clinical Trials, Inc., Altamonte Springs, Florida
  - Clinical Therapeutics Corporation, Coral Gables, Florida
  - Florida Research Network, Llc, Gainesville, Florida
  - Fpa Clinical Research, Kissimmee, Florida
  - Nextphase Clinical Trials, Inc., Miami, Florida
  - Middle Georgia Drug Study Center, Llc, Perry, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - Deerbrook Medical Associates, Vernon Hills, Illinois
  - Jackson Clinic, Rolling Fork, Mississippi
  - Mercy Medical Group/Dba Woodlake Research, Chesterfield, Missouri
  - Hudson Valley Clinical Research Center, Kingston, New York
  - Metrolina Medical Research, Charlotte, North Carolina
  - Crescent Medical Research, Salisbury, North Carolina
  - Community Health Care, Inc., Canal Fulton, Ohio
  - Wells Institute For Health Awareness, Kettering, Ohio
  - Newark Physician Associates, Newark, Ohio
  - Physician Research, Inc., Zanesville, Ohio
  - Gilbert Medical Research, Llc, Bethany, Oklahoma
  - Integris Family Care South Penn, Oklahoma City, Oklahoma
  - Integris Family Care Yukon, Yukon, Oklahoma
  - Willamette Valley Clinical Studies, Eugene, Oregon
  - Commonwealth Primary Care, Pc / Fleetwood Clinical Research, Fleetwood, Pennsylvania
  - Biomedical Research Associates, Llc, Shippensburg, Pennsylvania
  - Safe Harbor Clinical Research, East Providence, Rhode Island
  - Southeastern Research Associates, Inc., Greenville, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Middle Tennessee Clinical Research, Fayetteville, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Endocrine Associates, Houston, Texas
  - Village Family Practice, Houston, Texas
  - Non-Invasive Cardiovascular, Pa, Houston, Texas
  - Excel Clinical Research, Llc, Houston, Texas
  - Texas Center For Drug Development, Houston, Texas
  - Inst. Of Clin. Research At The Diabetes Cntr. Of The Sw, Midland, Texas
  - Hill Country Medical Associates, New Braunfels, Texas
  - Southwest Clinical Research Center, Llc, Pearland, Texas
  - Covenant Clinical Research, Pa, San Antonio, Texas
  - S.A.M. Clinical Research Center, San Antonio, Texas
- Mexico (11):
  - Local Institution, Pachuca, Hidelgo
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Morelia, Michioacan
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Monterrey, Nl, Nuevo León
  - Local Institution, Tampico, Tamaulipas
  - Local Institution, Mérida, Yucatán
  - Local Institution, Aguascalientes
  - Local Institution, Durango
  - Local Institution, Veracruz
- Philippines (6):
  - Local Institution, Cebu City
  - Local Institution, Jaro Iloilo City
  - Local Institution, Las Piñas
  - Local Institution, Marikina City
  - Local Institution, Pasig
  - Local Institution, Quezon City
- Puerto Rico (3):
  - Local Institution, Villa Fontana, Carolina
  - Local Institution, Ponce
  - Local Institution, San Juan
- Russia (12):
  - Local Institution, Arkhangelsk
  - Local Institution, Dzerzhinskiy
  - Local Institution, Kemerovo
  - Local Institution, Moscov
  - Local Institution, Moscow
  - Local Institution, Nizhny Novgorod
  - Local Institution, Novosibirsk
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov
  - Local Institution, Volgograd
  - Local Institution, Voronezh
  - Local Institution, Yaroslav
- South Korea (6):
  - Local Institution, Guri-si, Gyeonggi-do
  - Local Institution, Seoul, Nowon-Gu
  - Local Institution, Bucheon-si
  - Local Institution, Incheon
  - Local Institution, Seoul
  - Local Institution, Sungnam-Si, Gyeonggi-Do
- Ukraine (7):
  - Local Institution, Dnipro
  - Local Institution, Donetsk
  - Local Institution, Kiev
  - Local Institution, Lviv
  - Local Institution, Odesa
  - Local Institution, Vinnytsia
  - Local Institution, Zhytomyr

REFERENCES:
- [Result] Henry RR, Murray AV, Marmolejo MH, Hennicken D, Ptaszynska A, List JF. Dapagliflozin, metformin XR, or both: initial pharmacotherapy for type 2 diabetes, a randomised controlled trial. Int J Clin Pract. 2012 May;66(5):446-56. doi: 10.1111/j.1742-1241.2012.02911.x. Epub 2012 Mar 13. PMID 22413962
- [Derived] Kohan DE, Fioretto P, Johnsson K, Parikh S, Ptaszynska A, Ying L. The effect of dapagliflozin on renal function in patients with type 2 diabetes. J Nephrol. 2016 Jun;29(3):391-400. doi: 10.1007/s40620-016-0261-1. Epub 2016 Feb 19. PMID 26894924
- See also: Publication — http://onlinelibrary.wiley.com/doi/10.1111/j.1742-1241.2012.02911.x/epdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 994 participants enrolled, 632 completed a qualification period. Of these 632 participants, 603 were randomized. Of these 603 randomized, 598 received at least one dose of study medication treatment. Of these 598 randomized, 518 completed double-blind treatment period.
Groups:
- Dapagliflozin 5 mg + Metformin XR: Dapagliflozin tablets, oral, once daily for 24 weeks plus metfomin XR tablets (up to 2000mg), oral, once daily for 24 weeks
- Dapagliflozin 5 mg: Dapagliflozin tablets, oral, once daily for 24 weeks
- Metformin XR: Metfomin XR tablets (500mg up to 2000mg), oral, once daily for 24 weeks
Period: Overall Study
Arm/Group | Dapagliflozin 5 mg + Metformin XR | Dapagliflozin 5 mg | Metformin XR
Started | 194 | 203 | 201
Completed | 177 | 170 | 171
Not Completed | 17 | 33 | 30
Not completed — Death | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Adverse Event | 2 | 6 | 6
Not completed — Lost to Follow-up | 4 | 6 | 9
Not completed — Withdrawal by Subject | 8 | 15 | 9
Not completed — Non-compl., not met criteria, etc. | 3 | 4 | 6

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 5 mg + Metformin XR | Dapagliflozin 5 mg | Metformin XR | Total
Number analyzed (Participants) | 194 | 203 | 201 | 598
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.7 (9.31) | 52.3 (10.20) | 51.8 (9.80) | 52.0 (9.77)
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 177 | 183 | 184 | 544
  65 to younger than 75 years | 17 | 17 | 16 | 50
  75 years and older | 0 | 3 | 1 | 4
Sex/Gender, Customized [Number; unit: Participants]
  Male | 78 | 92 | 95 | 265
  Female | 116 | 111 | 106 | 333
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 153 | 166 | 158 | 477
  Black/African American | 8 | 4 | 6 | 18
  Asian | 32 | 33 | 35 | 100
  Other | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1C (HbA1c) at Week 24 (Last Observation Carried Forward [LOCF])
Description: HbA1c was measured as percent of hemoglobin by a central laboratory. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. HbA1c measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 4, 8, 12, 16, 20, and 24 in the double- blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: % of hemoglobin
Arm/Group | Dapagliflozin 5 mg + Metformin XR | Dapagliflozin 5 mg | Metformin XR
Number analyzed (Participants) | 185 | 196 | 195
% of hemoglobin | -2.05 (0.0892) | -1.19 (0.0866) | -1.35 (0.0868)
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg + Metformin XR vs Dapagliflozin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Primary endpoint was tested at alpha=0.05; significance was claimed only if DAPA 5MG + MET was superior to both controls; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-1.11 to -0.62], Standard Error of Mean 0.1243
Statistical Analysis 2: Comparison: Dapagliflozin 5 mg + Metformin XR vs Metformin XR; Test type: Superiority or Other; p < 0.0001, ANCOVA — Primary endpoint was tested at alpha=0.05; significance was claimed only if DAPA 5MG + MET is superior to both controls; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-0.94 to -0.45], Standard Error of Mean 0.1245

2. Secondary Outcome: Adjusted Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Fasting plasma glucose was measured as milligrams per deciliter(mg/dL) by a central laboratory. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. FPG measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24 in the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing FPG values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Dapagliflozin 5 mg + Metformin XR | Dapagliflozin 5 mg | Metformin XR
Number analyzed (Participants) | 192 | 203 | 200
mg/dL | -61.0 (2.783) | -42.0 (2.708) | -33.6 (2.728)
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg + Metformin XR vs Dapagliflozin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05. Significance was claimed only if DAPA 5MG + MET is superior to both controls; Mean Difference (Final Values) = -19.1, 95% CI 2-sided [-26.7 to -11.4], Standard Error of Mean 3.883
Statistical Analysis 2: Comparison: Dapagliflozin 5 mg + Metformin XR vs Metformin XR; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -27.5, 95% CI 2-sided [-35.1 to -19.8], Standard Error of Mean 3.897

3. Secondary Outcome: Percentage of Participants Achieving a Therapeutic Glycemic Response (Hemoglobin A1c [HbA1C]) <7.0% at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Percent adjusted for baseline HbA1c. Therapeutic glycemic response is defined as HbA1c <7.0%. Data after rescue medication was excluded from this analysis. HbA1c was measured as a percent of hemoglobin. Mean and standard error for percentage of participants estimated by modified logistic regression model.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: Percentage of participants
Arm/Group | Dapagliflozin 5 mg + Metformin XR | Dapagliflozin 5 mg | Metformin XR
Number analyzed (Participants) | 185 | 196 | 195
Percentage of participants | 52.4 (3.581) | 22.5 (2.741) | 34.6 (3.296)
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg + Metformin XR vs Dapagliflozin 5 mg; Test type: Superiority or Other; p < 0.0001, modified logistic regression — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 29.9, 95% CI 2-sided [20.8 to 39.0], Standard Error of Mean 4.633
Statistical Analysis 2: Comparison: Dapagliflozin 5 mg + Metformin XR vs Metformin XR; Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 17.8, 95% CI 2-sided [8.1 to 27.4], Standard Error of Mean 4.947

4. Secondary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1C (HbA1c) in Subjects With Baseline HbA1c ≥ 9% at Week 24 (Last Observation Carried Forward [LOCF])
Description: HbA1c was measured as percent of hemoglobin by a central laboratory. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. HbA1c measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 4, 8, 12, 16, 20, and 24 in the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing values at baseline and Week 24 (LOCF) in subjects with baseline HbA1c ≥ 9%
Measure: Mean (Standard Error); unit: % of hemoglobin
Arm/Group | Dapagliflozin 5 mg + Metformin XR | Dapagliflozin 5 mg | Metformin XR
Number analyzed (Participants) | 92 | 96 | 101
% of hemoglobin | -3.01 (0.1381) | -1.67 (0.1361) | -1.82 (0.1320)
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg + Metformin XR vs Dapagliflozin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.34, 95% CI 2-sided [-1.72 to -0.96], Standard Error of Mean 0.1938
Statistical Analysis 2: Comparison: Dapagliflozin 5 mg + Metformin XR vs Metformin XR; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.19, 95% CI 2-sided [-1.57 to -0.82], Standard Error of Mean 0.1912

5. Secondary Outcome: Adjusted Mean Change From Baseline in Total Body Weight (kg) at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Adjusted mean change from baseline in total body weight at Week 24 (or the last postbaseline measurement prior to Week 24 if no Week 24 assessment was available was determined. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. Body weight measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24 of the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: kg
Arm/Group | Dapagliflozin 5 mg + Metformin XR | Dapagliflozin 5 mg | Metformin XR
Number analyzed (Participants) | 192 | 203 | 200
kg | -2.66 (0.2428) | -2.61 (0.2361) | -1.29 (0.2378)
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg + Metformin XR vs Dapagliflozin 5 mg; Test type: Superiority or Other; p = 0.8769, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.72 to 0.61], Standard Error of Mean 0.3388
Statistical Analysis 2: Comparison: Dapagliflozin 5 mg + Metformin XR vs Metformin XR; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.37, 95% CI 2-sided [-2.04 to -0.71], Standard Error of Mean 0.3399

6. Secondary Outcome: Adjusted Mean Change From Baseline in Total Body Weight (kg) in Subjects With Baseline Body Mass Index (BMI) ≥ 27 kg/m^2 at Week 24 (Last Observation Carried Forward [LOCF])
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing values at baseline and Week 24 (LOCF) in subjects with BMI ≥ 27 kg/m2
Measure: Mean (Standard Error); unit: kg
Arm/Group | Dapagliflozin 5 mg + Metformin XR | Dapagliflozin 5 mg | Metformin XR
Number analyzed (Participants) | 142 | 156 | 154
kg | -3.04 (0.3031) | -2.88 (0.2890) | -1.47 (0.2907)
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg + Metformin XR vs Dapagliflozin 5 mg; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.98 to 0.66], Standard Error of Mean 0.4191
Statistical Analysis 2: Comparison: Dapagliflozin 5 mg + Metformin XR vs Metformin XR; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.57, 95% CI 2-sided [-2.40 to -0.74], Standard Error of Mean 0.4201

ADVERSE EVENTS:
Time Frame: Onset on or after the first date of double-blind treatment and on or prior to the last day of double-blind treatment 24 weeks plus 4 days for non-serious adverse event; plus 30 days for serious adverse event.
Arm/Group | Dapagliflozin 5 mg + Metformin XR | Dapagliflozin 5 mg | Metformin XR
Serious Adverse Events (participants affected / at risk) | 6/194 | 9/203 | 7/201
Other Adverse Events (participants affected / at risk) | 48/194 | 32/203 | 40/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 5 mg + Metformin XR (N=194) | Dapagliflozin 5 mg (N=203) | Metformin XR (N=201)
PULMONARY TUBERCULOSIS (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GANGRENE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OESOPHAGITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ISCHAEMIC NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 5 mg + Metformin XR (N=194) | Dapagliflozin 5 mg (N=203) | Metformin XR (N=201)
DIARRHOEA (Gastrointestinal disorders) | 15 (20) | 8 (9) | 14 (21)
NAUSEA (Gastrointestinal disorders) | 11 (20) | 4 (5) | 8 (14)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 (11) | 10 (11) | 11 (11)
URINARY TRACT INFECTION (Infections and infestations) | 10 (11) | 9 (9) | 10 (12)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 9 (9) | 11 (13) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No